CLINICAL TRIAL: NCT06939712
Title: A Study on the Impact of Online Positive Psychological Intervention on the Mental Health and Quality of Life of Crohn's Disease Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang University (Other); Shaoxing Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024-0629IR2024327
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Positive Psychology Intervention Group (Experimental): Intervention group patients will participate in a 6-week online psychological support program, held once a week. The sessions will primarily be organized by a facilitator and will include patient-led discussions and communication. The specialized nurse will add the patients to the corresponding WeChat group and collect general information about the research subjects. A nursing graduate student (blinded) will collect data before the intervention, at the end of the third week of the intervention, at the end of the sixth week of the intervention, and three months after the end of the intervention. Five group leaders, all trained in a standardized manner, will carry out interventions according to the intervention plan and content for the patients in the intervention group. IBD specialists and nurses will implement routine patient management.
  Interventions: Behavioral: Online Positive Psychology Intervention
- Routine Care Group (Placebo Comparator): The IBD specialists and nurses will primarily provide health education on IBD disease knowledge, medication, diet, exercise, lifestyle, psychological well-being, and follow-up care based on the patient's actual situation and individual needs during patient follow-up visits. At the same time, patients will be added to the control group WeChat group.
  Interventions: Other: Routine Care

INTERVENTIONS:
Behavioral: Online Positive Psychology Intervention — A 6-week online psychological support program, held once a week, primarily organized by a facilitator, with patient-led discussions and communication.
  Arms: Online Positive Psychology Intervention Group
Other: Routine Care — A 6-week program of health education provided by IBD specialists and nurses during patient follow-ups, tailored to individual patient circumstances and needs. Topics include IBD disease knowledge, medication management, diet, exercise, lifestyle, psychological support, and follow-up care. Patients in this group will also join a control group WeChat group for study-related communication.
  Arms: Routine Care Group

SUMMARY:
Crohn's disease (CD) is a chronic, nonspecific inflammatory disease that can affect the entire digestive tract. It is difficult to cure and often relapses, causing long-term suffering for patients. This persistent condition significantly impacts their mental and psychological well-being, leading to a noticeable decline in their quality of life. Furthermore, these negative emotions can contribute to disease recurrence and the worsening of symptoms. Positive psychological intervention (PPI) refers to the enhancement of positive emotions, cognition, and behaviors to increase well-being and alleviate symptoms. Therefore, this study aims to use psychological methods to help CD patients better recognize and understand their positive experiences, thus aiding them in coping with stress and adversity more effectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Crohn's disease according to the 2018 diagnostic criteria established by the Inflammatory Bowel Disease Group of the Chinese Medical Association's Gastroenterology Branch;
* Patients aged between 18 and 75 years;
* Patients with a score of 5-14 on the GAD-7 (indicative of mild to moderate anxiety) or a score of 5-14 on the PHQ-9 (indicative of mild to moderate depression);
* Patients who understand and agree to comply with the study requirements and have signed informed consent;
* Patients who are able to read and access the internet, either independently or with assistance from a family member, and are capable of using WeChat and mobile applications;
* Patients who are able to complete all course trainings and/or follow-up procedures.

Exclusion Criteria:

* Individuals with a history or current diagnosis of psychiatric illness or cognitive impairment, or those currently taking psychiatric medications; Individuals working in the field of psychology, or those who have previously studied or are currently studying positive psychology;
* Individuals with concurrent other intestinal diseases or malignancies;
* Individuals with severe primary diseases of the cardiovascular, cerebrovascular, hepatic, or renal systems.

Withdrawal Criteria:

* Patients lost to follow-up due to withdrawal or other reasons during the intervention period;
* Patients who develop severe complications or experience significant changes in their condition that prevent them from continuing the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
GAD-7 | Measurements will be conducted at four time points: prior to the intervention, at the end of Week 3 of the intervention, at the end of Week 6 of the intervention, and three months after the intervention concludes.
  indicative of mild to moderate anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Hangzhou, Zhejiang, China